CLINICAL TRIAL: NCT07385768
Title: The Effect of an Eye Mask-Based Blackout Protocol on Patients' Sleep Quality and Melatonin Levels: A Randomised Controlled Trial
Brief Title: Effect of an Eye Mask-Based Blackout Protocol on Sleep Quality and Melatonin
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ataturk University (Other)
Responsible Party: Principal Investigator, Bahar Ciftci, Principal Investigator, Ataturk University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ATAUNI-SLEEP-ICU-01
Record Dates: First submitted 2026-01-20; First posted 2026-02-04 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-01

CONDITIONS: Sleep Disturbance; Circadian Rhythm Sleep Disorders; Intensive Care Unit Patients
Keywords: Eye mask; Light exposure; Melatonin; Sleep quality; Intensive care unit
MeSH Terms: conditions — Parasomnias; Sleep Disorders, Circadian Rhythm; Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Intervention Model Description: Participants were randomly assigned to either an intervention group or a control group and followed in parallel throughout the study period.
Who Masked: Investigator, Outcomes Assessor
Masking Description: Laboratory personnel analysing urinary melatonin levels and the statistician performing data analysis were blinded to group allocation. Due to the nature of the intervention, participants and bedside nurses could not be blinded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Eye Mask Intervention Group (Experimental): Participants received a nighttime eye mask-based blackout protocol during sleep hours in the intensive care unit in addition to routine care.
  Interventions: Other: Eye Mask-Based Blackout Protocol
- Control Group (No Intervention): Participants received routine intensive care without the use of an eye mask.

INTERVENTIONS:
Other: Eye Mask-Based Blackout Protocol — A non-pharmacological nursing intervention involving the use of an eye mask during nighttime sleep to reduce light exposure and support circadian rhythm regulation in intensive care unit patients.
  Arms: Eye Mask Intervention Group

SUMMARY:
Sleep disturbance is a common problem among patients hospitalized in intensive care units due to continuous light exposure, noise, and frequent medical interventions. Disruption of the normal day-night cycle may reduce melatonin secretion and negatively affect sleep quality and recovery.

This randomized controlled study aimed to evaluate the effect of an eye mask-based blackout protocol on sleep quality and melatonin levels in patients hospitalized in a chest intensive care unit. Participants were randomly assigned to either an intervention group or a control group. Patients in the intervention group wore a lightproof eye mask during nighttime hours (11:00 p.m. to 05:00 a.m.) in addition to standard light-reduction practices, while the control group received routine intensive care.

Sleep quality was assessed using validated subjective scales, and melatonin levels were evaluated by measuring urinary 6-sulfatoxymelatonin. The study sought to determine whether reducing nighttime light exposure using a simple, non-invasive intervention could improve sleep quality and support circadian rhythm regulation in intensive care patients.

DETAILED DESCRIPTION:
This study was designed as a randomized controlled trial to investigate the effect of an eye mask-based blackout protocol on sleep quality and melatonin levels in patients hospitalized in a chest intensive care unit.

The study was conducted at a university research hospital in Turkey. Eligible adult patients who were conscious, breathing spontaneously, and able to provide informed consent were randomly assigned to either an intervention group or a control group using a 1:1 allocation ratio. Patients receiving mechanical ventilation or using medications affecting melatonin secretion were excluded.

Participants in the intervention group wore a lightproof eye mask between 11:00 p.m. and 05:00 a.m. for two consecutive nights. In addition to eye mask use, nighttime lighting in the patient's room was minimized according to a standardized protocol. The control group received routine intensive care without any additional light-reduction intervention.

Sleep quality was evaluated using the Visual Analogue Scale for Sleep Quality and the Richard Campbell Sleep Scale. Melatonin secretion was assessed by measuring urinary 6-sulfatoxymelatonin levels collected overnight. Urine samples were stored under controlled conditions and analyzed using an enzyme-linked immunosorbent assay (ELISA).

The primary objective of the study was to determine whether the eye mask-based blackout protocol improved subjective sleep quality. A secondary objective was to assess changes in melatonin levels as a biological marker of circadian rhythm regulation.

All procedures were conducted in accordance with the Declaration of Helsinki. Ethical approval was obtained from the relevant institutional ethics committee, and written informed consent was obtained from all participants prior to enrollment.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients aged 18 years and older
* Patients admitted to the intensive care unit
* Patients expected to remain in the intensive care unit for at least 24 hours
* Patients with the ability to tolerate an eye mask during nighttime sleep
* Patients or their legal representatives who provided informed consent

Exclusion Criteria:

* Patients with facial trauma, eye injury, or ophthalmologic conditions preventing eye mask use
* Patients receiving continuous deep sedation
* Patients with severe cognitive impairment or delirium preventing cooperation
* Patients with diagnosed sleep disorders prior to intensive care admission
* Patients who refused to participate in the study

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2024-08-01 (Actual); Primary Completion 2025-05-01 (Actual); Study Completion 2025-06-01 (Actual)

PRIMARY OUTCOMES:
Sleep quality (Richard-Campbell Sleep Questionnaire [RCSQ] total score) | Measured twice: (1) baseline-morning of ICU day 2 (after the first night, 23:00-05:00), and (2) post-intervention-morning of ICU day 3 (after the blackout night with eye mask from 23:00 to 05:00).
  Change in sleep quality assessed using the Richard-Campbell Sleep Questionnaire (6 items, 0-100 VAS each; higher scores indicate better sleep). The total score is calculated as the mean of all item scores.

SECONDARY OUTCOMES:
Sleep quality (Visual Analogue Scale [VAS], 1-10) | Measured twice: (1) baseline-morning of ICU day 2 (after the first night, 23:00-05:00), and (2) post-intervention-morning of ICU day 3 (after the blackout night with eye mask from 23:00 to 05:00).
  Self-reported sleep quality rated on a 1-10 scale (1 = worst sleep quality, 10 = best sleep quality).
Urinary 6-sulfatoxymelatonin (aMT6s) level (ng/mg creatinine) | Measured twice using overnight urine collection: (1) baseline-urine accumulated from 23:00 to 05:00 on the first night (ICU day 2 morning sample), and (2) post-intervention-urine accumulated from 23:00 to 05:00 on the blackout night with eye mask (ICU da
  Change in melatonin secretion assessed by urinary 6-sulfatoxymelatonin (aMT6s) measured by ELISA and normalized to urinary creatinine (ng/mg creatinine). Urine was collected via Foley catheter drainage.

CONTACTS AND LOCATIONS:
Locations (1):
- Atatürk University Faculty of Nursing, Erzurum, Erzurum, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No